CLINICAL TRIAL: NCT05242536
Title: The Effect of a Nurse-led Program on Psychosocial Problems and Quality of Life in Stroke Patients
Brief Title: A Nurse-led Program for Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Istinye University (Other)
Responsible Party: Principal Investigator, Zeliha Tülek, Assoc.Prof, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Nurse-led Program for Stroke
Record Dates: First submitted 2022-01-23; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Stroke; Psychosocial Problems
Keywords: Stroke; Psychosocial Problem; Nurse-led Program; Quality of Life
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse- led program (Experimental): A nurse coordinated multidisciplinary program aiming to improve psychosocial problems has been developed and will be applied to the patients in the experimental group. This nurse-led program will start at discharge and continue for three months.
  Interventions: Other: Nurse- led program
- Routine follow-up group (No Intervention): The control group will be applied usual care. Patients in the control group will be discharged by receiving standard care and performing discharge trainings used in the routine care.

INTERVENTIONS:
Other: Nurse- led program — A nurse coordinated multidisciplinary program aiming to improve psychosocial problems has been developed and will be applied to the patients in the experimental group. This nurse-led program will start at discharge and continue for three months.
  Arms: Nurse- led program

SUMMARY:
The aim of this study is to examine the effectiveness of nurse- led program on psychosocial problems and quality of life in stroke patients. This randomized controlled trial will be conducted in Stroke Center in Istinye University Liv Hospital-Bahcesehir. Eligible participants will be randomly allocated to either the control group (receiving usual care/ routine follow-up group) or the intervention group (receiving nurse-led psychosocial program). A nurse- led program will be implemented for the management of psychosocial problems following a comprehensive evaluation. Then, the effect of this program on psychosocial problems and quality of life will be evaluated in the 1st and 3rd months after discharge.

DETAILED DESCRIPTION:
The aim of this study is to examine the effectiveness of nurse- led program on psychosocial problems and quality of life in stroke patients. This randomized controlled trial will be conducted in Stroke Center in Istinye University Liv Hospital- Bahcesehir. Patients who meet the criteria will be randomized into the intervention group or control group. All patients will be assessed at discharge by use of following tools: National Institutes of Health Stroke Scale (NIHSS), modified Rankin Scale, Functional Independence Measure (FIM), Montreal Cognitive Assessment (MoCA), Hospital Anxiety and Depression Scale (HADS), Pittsburgh Sleep Quality Index (PSQI). A nurse coordinated multidisciplinary program aiming to improve psychosocial problems has been developed and will be applied to the patients in the experimental group. This nurse-led program will start at discharge and continue for three months. The control group will be applied usual care. Two groups will be compared at baseline and at the 3rd month after discharge in terms of psychosocial variables and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Be literate
* Have a clinical diagnosis of ischemic stroke
* History of any preceding cerebral vascular event
* Capable of giving informed consent

Exclusion Criteria:

* Age ≤ 18 years
* Have a mental disorder that will prevent cognitive evaluation
* Have an impaired consciousness (confusion, delirium, etc.)
* History of any type of cognitive decline
* Have severe neurologicial deficit
* Severe aphasia
* Living in a nursing home
* Known malignant disease or other chronic disease with poor prognosis and a low life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Montreal Cognitive Assessment Test scores | At the baseline, 1st and 3rd month after discharge
  Cognitive function will be evaluated by Montreal Cognitive Assessment Test.
Change in Hospital Anxiety and Depression Scale scores | At the baseline, 1st and 3rd month after discharge
  Anxiety and depression will be evaluated by Hospital Anxiety and Depression Scale.
Change in Pittsburgh Sleep Quality Index scores | At the baseline, 1st and 3rd month after discharge
  Sleep quality will be evaluated by Pittsburgh Sleep Quality Index.

SECONDARY OUTCOMES:
Change in Fatigue Severity Scale scores | At the 1st and 3rd month after discharge
  Fatigue will be evaluated by Fatigue Severity Scale.
Change in Reintegration to Normal Living Index scores | At the 1st and 3rd month after discharge
  Adaptation to life will be evaluated by Reintegration to Normal Living Index.
Change in Stroke Specific Quality of Life Scale scores | At the 1st and 3rd month after discharge
  Quality of life will be evaluated by Stroke Specific Quality of Life Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Hilalnur Kucukakgun, RN,MSc, Principal Investigator — Istanbul University - Cerrahpasa; Zeliha Tulek, RN,Assoc Prof, Study Director — Istanbul University - Cerrahpasa; Yakup Krespi, MD, Prof, Study Chair — Istinye University Liv Hospital- Bahcesehir
Locations (1):
- Stroke Center in Istinye University Liv Hospital-Bahcesehir, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verberne DPJ, Kroese MEAL, Staals J, Ponds RWHM, van Heugten CM. Nurse-led stroke aftercare addressing long-term psychosocial outcome: a comparison to care-as-usual. Disabil Rehabil. 2022 Jun;44(12):2849-2857. doi: 10.1080/09638288.2020.1849417. Epub 2020 Nov 26. PMID 33242261
- [Result] Lanctot KL, Lindsay MP, Smith EE, Sahlas DJ, Foley N, Gubitz G, Austin M, Ball K, Bhogal S, Blake T, Herrmann N, Hogan D, Khan A, Longman S, King A, Leonard C, Shoniker T, Taylor T, Teed M, de Jong A, Mountain A, Casaubon LK, Dowlatshahi D, Swartz RH; Management of Mood, Cognition and Fatigue Following Stroke Best Practice Writing Group, the Heart & Stroke Canadian Stroke Best Practices and Quality Advisory Committee; in collaboration with the Canadian Stroke Consortium. Canadian Stroke Best Practice Recommendations: Mood, Cognition and Fatigue following Stroke, 6th edition update 2019. Int J Stroke. 2020 Aug;15(6):668-688. doi: 10.1177/1747493019847334. Epub 2019 Jun 21. PMID 31221036